CLINICAL TRIAL: NCT00844896
Title: RCT Intervention to Reduce Stress in 0-5 Year Olds With Burns
Brief Title: Intervention to Reduce Stress in 0-5 Year Olds With Burns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Frederick J. Stoddard, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: SHC Grant No. 8894
Record Dates: First submitted 2009-02-12; First posted 2009-02-16 (Estimated); Results first posted 2014-10-16 (Estimated); Last update posted 2014-10-16 (Estimated); Status verified 2014-10

CONDITIONS: Stress, Psychological; Post-Traumatic Stress Disorder; Major Injury
Keywords: Pathological stress & PTSD in preschool children & parents; Child and parent resilience after burn trauma
MeSH Terms: conditions — Stress, Psychological; Stress Disorders, Post-Traumatic | interventions — Psychosocial Intervention; butyl phosphorotrithioate

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- DEF-only (Active Comparator): Distress Emotional Support and Family Assessment Treatment
  Interventions: Behavioral: DEF-only
- DEF + COPE (Experimental): Distress Emotional Support and Family Assessment Treatment and Creating Opportunities for Parent Empowerment Treatment
  Interventions: Behavioral: DEF + COPE

INTERVENTIONS:
Behavioral: DEF-only — The DEF protocol is from the National Child Traumatic Stress Network (NCTSN). DEF provides a sequential methodology for clinicians to assess medically traumatized children and their families and to plan specific interventions for them.
  In the present study, the DEF intervention is both a generalized approach taught to all Shriners Hospitals for Children (SHC)- Boston clinical staff, and for those participants of the present study, consists of an optional meeting with a member of the SHC Psychiatry Department. During this meeting, parents will have the chance to review any areas of pain, anxiety, or support that came up during their interviews or any other areas of concern about their child or his/her hospitalization that they wish to raise.
  Other Names: Psychosocial Intervention
  Arms: DEF-only
Behavioral: DEF + COPE — All enrolled participants will be offered the chance to meet with a psychiatric clinician for the DEF component of the intervention.
  For those assigned to receive COPE (Creating Opportunities for Parent Empowerment), parents will receive one of two versions of the materials: one for children less than one year old, and one for children ages 1-5 years. The COPE program was adapted for children with burns and developed to target major stressors that parents experience when their children are hospitalized, such as the loss of parental control. COPE also contains a behavioral component to help parents to carry out the recommendations provided to them. Each of these versions of the COPE program is essentially self-administered to parents via audio tapes and activity workbooks.
  Other Names: Psychosocial Intervention
  Arms: DEF + COPE

SUMMARY:
The objectives of this study are to test and validate a simple, feasible intervention to reduce pediatric burn traumatic stress in 0-5 year old children and their parents.

We have refined and implemented an early post-burn psychosocial assessment and intervention for stress reduction for young children and their parents based on the "DEF" Protocol (Distress, Emotional Support, Family) from NCTSN's 'Pediatric Medical Toolkit for Health Care Providers,' and a burn specific version of the COPE (Creating Opportunities for Parent Empowerment)intervention.

It is hypothesized that the combined DEF + COPE Intervention will be simple to implement and use under both experimental and real world conditions. The proof of the latter hypothesis will be that staff at Shriners Hospitals for Children-Boston will willingly incorporate it into routine care by the end of the project.

We will evaluate, using an RCT design, the DEF + COPE Intervention by comparing outcomes for subjects who are randomly assigned to receive it with outcomes for subjects who are assigned to receive the DEF Intervention only.

It is hypothesized that children in the DEF + COPE Intervention Group will show significantly greater decreases over time in pain and anxiety ratings, heart rate, PTSD total symptom scores and physiological symptom scores (such as heart rate and heart rate variability from baseline to follow up) than will children in the DEF-only group. Similarly, it is hypothesized that parents assigned to the DEF + COPE group will show significantly decreased scores on the Stanford PTSD measure.

DETAILED DESCRIPTION:
Despite their clear vulnerability and demonstrated need, preschool children and their families have been the subject of very little research on traumatic stress following all types of injuries including burns (Stoddard & Saxe, 2001). This lack of research is even more critical in an age in which tragic and traumatic events are increasing in frequency and severity.

Early identification of young burn survivors who also have elevated heart rates, high levels of pain and/or exhibit other symptoms of PTSD may help to prevent the development of later psychopathology. If assessment of stress is improved, then early interventions may be designed to prevent or reduce the later emergence of PTSD including phobias and associated symptoms. As of this time, however, no early interventions are available for very young burned children.

The intervention is driven by the findings of our previous study of 1-4 year olds that suggested that the child's PTSD symptoms could be reduced by improved pain and anxiety control and by reduced parental PTSD. The current study aims to advance the science of prevention of pathological stress responses in preschool children and their parents, strengthen both child and parent resilience after burn trauma and its treatments, and provide interventions for the children with posttraumatic symptoms such as re-experiencing, hyperarousal, avoidance, insomnia, nightmares, or regressions in social abilities like smiling and/or vocalization.

Our goal is not only to set up an intervention that will be effective in reducing stress for young children with burns and their families, we also want to assure that the intervention is feasible and sustainable for implementation in Shriners Hospital Boston, other Shriners Hospitals, and other Level I Pediatric Burn Centers after the end of this project.

The models for intervention are:

- COPE (Creating Opportunities for Parent Empowerment)

The psychosocial intervention which holds the greatest promise as a treatment for young burned children and their families is the COPE (Creating Opportunities for Parent Empowerment) program. COPE was designed to be implemented in a tertiary care center with seriously ill children. It has been shown in more than a dozen studies to significantly reduce symptoms of stress in both children and their parents. In one study, Melnyk et al (2004) delivered the COPE program with audiotapes and matching written information, and a parent-child workbook that helped implement the audiotaped information. It focused on increasing: 1) parents' knowledge and understanding the range of behaviors and emotions that young children typically display during and after hospitalization and 2) direct parent participation in their children's' emotional and physical care. In collaboration with COPE's senior author, B. M. Melnyk, the COPE intervention and materials will be tailored for a population of young burned children at Shriners Hospitals for Children-Boston.

Melnyk and her colleagues (2004; 1997; 2006) developed COPE as a "theory-based educational-behavioral program that consists of two types of educational information: (a) child behavioral information that teaches parents about the most typical emotions and behavioral responses that young children manifest as they cope with illness or trauma and hospitalization, and (b) parental role information that provides parents with suggestions regarding how they can best help their children to cope with the hospital experience" (Melnyk, Feinstein, Alpert-Gillis et al., 2006, p. 475). The COPE program was developed to target two major stressors that parents experience when their children are hospitalized: 1) their children's emotions, behaviors, and physical characteristics and 2) the loss of the parental role/control. COPE also contains a behavioral component to help parents to carry out the recommendations provided to them in the educational information.

There are now three versions of the COPE program: (a) COPE for parents of young hospitalized children, 1 to 7 years of age, (b) COPE: PICU for parents of 2 to 7-year- old critically ill young children, and (c) COPE: NICU for parents of low-birth-weight (LBW) premature infants. Each of these versions of the COPE program is essentially self-administered to parents via audio tapes and activity workbooks, generally in three brief (15 minute) sessions over a two day period during a pediatric hospitalization. Examples of workbook activities are teaching their children about how to express their feelings through play with their children and reading the Jenny's Wish book (i.e., a story about a small child who copes successfully with a critical care hospitalization). The suggested administration times are: 6-16 hours after admission to PICU, 2-16 hours after transfer to general pediatric unit, and 2-3 days after discharge from hospital.

Multiple studies have shown the validity of COPE (Melnyk, 1994, 1995; Melnyk et al., 2004; Melnyk et al., 2001; Melnyk et al., 1997; Melnyk, Feinstein, & Fairbanks, 2006; Melnyk & Feinstein, 2001; Melnyk, Feinstein, Alpert-Gillis et al., 2006; Vulcan & Nikulich-Barrett, 1988). The 2004 paper describes an RCT design with 174 mother-child dyads that showed significant reductions in parental and child symptoms of stress at six and twelve months after the intervention.

- The Pediatric Medical Traumatic Stress Toolkit for Health Care Providers

The Pediatric Medical Traumatic Stress Toolkit for Health Care Providers provides another way to reduce unnecessary stress in medically ill children. Created by the National Child Traumatic Stress Network ("National Child Traumatic Stress Network (NCTSN) Toolkit for Health Care Providers,"; Stuber, Schneider, Kassam-Adams, Kazak, & Saxe, 2006), the Toolkit is another innovation that could provide a platform not only for identifying children and families who are most in need of the COPE intervention but also for interventions not addressed by COPE like finding additional parental support, providing additional pain, anxiety, or depression medication for children or parents, or designing more targeted interventions for children and families whose stress levels may be lower overall but high only in certain areas.

The Toolkit contains a protocol called 'D-E-F' that helps clinicians to assess medically traumatized children and their families and to plan specific interventions for them. The idea of the Toolkit is that after the standard ABC's (Airways, Breathing, Circulation) of medical problems have been dealt with, clinicians should attend to the next most important issues, the 'DEF's of problems. The DEF acronym stands for Distress, Emotional Support, and Family Functioning. As described later in this proposal, the DEF protocol will be the basis for the initial assessment and clinical intervention recommendations provided by child psychiatry staff as part of a new program being developed at SBH Boston. The Toolkit contains handouts to help parents understand the stresses their medically ill children are facing and to help their children to cope with them as well as an overarching framework for mental health and medical clinicians to use in assessing and intervening to minimize post traumatic stress reactions.

The Toolkit materials are designed primarily for hospital-based heath care providers like physicians and nurses, and for parents. The Toolkit promotes "trauma-informed practice of pediatric health care in hospital settings across the continuum of care… - e.g., from emergency care, to the ICU, to specialized inpatient units, to general pediatrics". The NCTSN Toolkit for Health Care Providers provides an overarching framework for healthcare workers to use for both assessment and intervention for PTSD in children and parents.

Working within the NCTSN, many medical and psychosocial professionals, including Drs. Saxe and Stoddard, spent several years formulating this approach to working with children who have injuries and medically related traumas (Stuber et al., 2006). The Toolkit was released in late 2004 and although it shows a great deal of promise, it has yet to be validated and applied as a part of routine clinical care. The proposed project will be the first to empirically test it as a part of an intervention strategy.

ELIGIBILITY:
Inclusion Criteria:

* All children between the ages of 0 to 5.9 years of age who are admitted to Shriners Hospitals for Children - Boston for an acute burn or reconstructive surgery
* Parent(s) or legal guardian is English- or Spanish-speaking
* Medical clinicians deem their patients appropriate candidates

Exclusion Criteria:

* Children whose primary physicians or nurses think that their patient or parent should not be approached for the study due to high levels of stress, criminal or child protective service involvement
* Children whose parents the Chief of Staff or his designee does not believe should be approached for study because they have not consented in general to a participation in research studies during their child's hospitalization
* Children who are so gravely ill that their parents do not wish to talk

The parents of initially excluded children may be approached for the study later in the child's hospital stay if any of these rule outs abate (most typically when a child is no longer critically ill).

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 57 (Actual)
Dates: Start 2008-05; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frederick J Stoddard Jr., MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Shriners Hospitals for Children, Boston, Massachusetts, United States

REFERENCES:
- [Background] Stoddard FJ, Saxe G, Ronfeldt H, Drake JE, Burns J, Edgren C, Sheridan R. Acute stress symptoms in young children with burns. J Am Acad Child Adolesc Psychiatry. 2006 Jan;45(1):87-93. doi: 10.1097/01.chi.0000184934.71917.3a. PMID 16327585
- [Background] Stoddard FJ, Ronfeldt H, Kagan J, Drake JE, Snidman N, Murphy JM, Saxe G, Burns J, Sheridan RL. Young burned children: the course of acute stress and physiological and behavioral responses. Am J Psychiatry. 2006 Jun;163(6):1084-90. doi: 10.1176/ajp.2006.163.6.1084. PMID 16741210
- [Background] Drake JE, Stoddard FJ Jr, Murphy JM, Ronfeldt H, Snidman N, Kagan J, Saxe G, Sheridan R. Trauma severity influences acute stress in young burned children. J Burn Care Res. 2006 Mar-Apr;27(2):174-82. doi: 10.1097/01.BCR.0000202618.51001.69. PMID 16566561
- [Background] Stuber ML, Schneider S, Kassam-Adams N, Kazak AE, Saxe G. The medical traumatic stress toolkit. CNS Spectr. 2006 Feb;11(2):137-42. doi: 10.1017/s1092852900010671. PMID 16520691
- [Background] Melnyk BM, Alpert-Gillis L, Feinstein NF, Crean HF, Johnson J, Fairbanks E, Small L, Rubenstein J, Slota M, Corbo-Richert B. Creating opportunities for parent empowerment: program effects on the mental health/coping outcomes of critically ill young children and their mothers. Pediatrics. 2004 Jun;113(6):e597-607. doi: 10.1542/peds.113.6.e597. PMID 15173543
- [Background] Stoddard FJ, Saxe G. Ten-year research review of physical injuries. J Am Acad Child Adolesc Psychiatry. 2001 Oct;40(10):1128-45. doi: 10.1097/00004583-200110000-00007. PMID 11589526

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Children aged 0-5 years who were hospitalized for an acute or reconstructive burn injury and their families were eligible for participation in the study. Recruitment for the study occurred from May 2008-August 2010.
Period: Overall Study
Arm/Group | DEF-only | DEF + COPE
Started | 29 | 28
Completed | 17 | 11
Not Completed | 12 | 17
Not completed — Lost to Follow-up | 12 | 16
Not completed — Parents did not have time to complete | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- DEF-only: 29 subjects in this arm of the study.
- DEF + COPE: 28 subjects in this arm of the study.
- Total: Total of all reporting groups
Arm/Group | DEF-only | DEF + COPE | Total
Number analyzed (Participants) | 29 | 28 | 57
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 29 | 28 | 57
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 1.9 (1.4) | 2.3 (1.6) | 2.1 (1.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 11 | 23
  Male | 17 | 17 | 34
Region of Enrollment [Number; unit: participants]
  United States | 29 | 28 | 57

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Burn Outcomes Questionnaire Short Form (0-4 Year Old Version) at Six Months
Description: Burn Outcomes Questionnaire (American Burn Association/Shriners Hospitals for Children) Short Form (0-4 year old version). Parent-rated questionnaire that focuses on child's pain and parent's worry. Scores range from 5-24, with a higher score indicative of worse outcomes. Change in scores was measured from baseline to six month follow-up
Time Frame: Baseline and six month follow-up
Population: Intention to Treat (ITT)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DEF-only | DEF + COPE
Number analyzed (Participants) | 13 | 6
units on a scale | -4.9 (4.6) | -4.5 (1.4)

2. Primary Outcome: Change From Baseline in Pediatric Symptom Checklist at Six Months
Description: Pediatric Symptom Checklist is an 18-item psychosocial checklist in which symptoms are rated from 0 (never) to 2 (often) and the last question is rated as yes or no (0 or 1). Items are summed and the score can range from 0-35, with a higher score indicative of more symptoms and a worse outcome. Change in scores were observed from baseline to six month follow-up
Time Frame: Baseline and six month follow-up
Population: Intention to Treat (ITT)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DEF-only | DEF + COPE
Number analyzed (Participants) | 5 | 2
units on a scale | 2.9 (7.9) | 1.0 (5.7)

3. Primary Outcome: Change From Baseline in Parenting Stress Index at Six Months
Description: Parenting Stress Index is a 12-item parent-rated questionnaire which employs a 1-5 Likert scale. Scores range from 12-60, with a lower score indicative of worse outcomes and a cutoff of 15. Change in scores were observed from baseline to six month follow-up.
Time Frame: Baseline and six month follow-up
Population: Intention to treat (ITT)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DEF-only | DEF + COPE
Number analyzed (Participants) | 10 | 4
units on a scale | 7.1 (12.6) | -3.3 (9.0)

4. Primary Outcome: Change From Baseline in Child Stress Reaction Checklist Short Form at Six Month
Description: Child Stress Reaction Checklist Short Form is a 9-item parent-rated checklist. Scores range from 0-18 with a higher score indicative of worse outcomes. Change in scores were observed from baseline to six month follow-up
Time Frame: Baseline and six month follow-up
Population: Intention to treat (ITT)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DEF-only | DEF + COPE
Number analyzed (Participants) | 15 | 7
units on a scale | 0.8 (2.5) | 0.7 (2.4)

5. Primary Outcome: Change From Baseline in PTSD Semi-Structured Interview at Six Months
Description: Posttraumatic Stress Disorder Semi-Structured Interview is based on DSM-IV criteria, with a higher score indicative of increased symptoms of PTSD. The total rating was scored from 19 questions in three clusters of symptoms, with a score range of 0-38. Change in scores were observed from baseline to six month follow-up.
Time Frame: Baseline and six-month follow-up
Population: Intention to treat (ITT)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DEF-only | DEF + COPE
Number analyzed (Participants) | 12 | 6
units on a scale | -1.7 (3.1) | -1.5 (4.6)

6. Primary Outcome: Change From Baseline in Hospital Emotional Support Form From Six Months
Description: Hospital Emotional Support Form is a 12-question form that rates parents/caregivers need for in-hospital emotional support. Scores range from 11-24, with a lower score indicative of worse outcomes. Change in scores were observed from baseline to six month follow-up.
Time Frame: Baseline and six-month follow-up
Population: Intention to treat (ITT)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DEF-only | DEF + COPE
Number analyzed (Participants) | 16 | 7
units on a scale | 1.1 (3.8) | 2.0 (2.6)

7. Primary Outcome: Change From Baseline in Stanford Acute Stress Reaction Questionnaire at Six Months
Description: Stanford Acute Stress Reaction Questionnaire is a 31-question self-report measure for acute stress in parents. Scores range from 0-155 with a higher score indicative of worse outcomes. Change in scores were observed from baseline to six month follow-up.
Time Frame: Baseline and six-month follow-up
Population: Intention to treat (ITT)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DEF-only | DEF + COPE
Number analyzed (Participants) | 14 | 6
units on a scale | -9.6 (42.5) | 13.8 (33.2)

8. Primary Outcome: DEF Participation
Description: Outcomes in this measure were quantified by the number of participants in either intervention (DEF-only or COPE+DEF). During the study, DEF intervention was part of the standard of care for all patients at Shriners Hospitals for Children-Boston and thus every participant in this study had been evaluated using DEF to determine distress, emotional and family support.
Time Frame: Baseline
Population: Intentional to treat (ITT)
Measure: Number; unit: participants
Arm/Group | DEF-only | DEF + COPE
Number analyzed (Participants) | 29 | 28
participants | 29 | 28

9. Primary Outcome: Change From Baseline in Burn Outcomes Questionnaire Short Form (5-18 Year Old Version) From Six Months.
Description: Burn Outcomes Questionnaire (American Burn Association/Shriners Hospitals for Children) Short Form (5-18 Year Old Version) is a 3-item questionnaire with scores ranging from 0-18. A higher score is indicative of worse outcomes. Used for five year olds in the study. Change in scores were observed from baseline to six month follow-up.
Time Frame: baseline and six month follow-up
Population: Intention to Treat (ITT)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DEF-only | DEF + COPE
Number analyzed (Participants) | 1 | 0
units on a scale | -0.2 (0.0) |

ADVERSE EVENTS:
Arm/Group | DEF-only | DEF + COPE
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/28
Other Adverse Events (participants affected / at risk) | 0/29 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No